CLINICAL TRIAL: NCT02731872
Title: The Effect of Oxygen Therapy With Airvo High-flow Heated Humidification for Respiratory Insufficiency in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: The Effect of Oxygen Therapy With Airvo High-flow Heated Humidification
Acronym: HHCOPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Birgitte Schantz Laursen (Other)
Collaborators: Fisher and Paykel Healthcare (Industry); AGA The Linde Group (Unknown)
Responsible Party: Sponsor-Investigator, Birgitte Schantz Laursen, Associated professor, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-20110057
Record Dates: First submitted 2016-03-14; First posted 2016-04-08 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: COPD
Keywords: COPD; oxygen treatment; quality of life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High Flow humidification system (Experimental): In addition to their usual oxygen apparatuses, the treatment group will have an Airvo humidifier system installed in the home. The supplied oxygen flow will be entrained along with room air through the Airvo humidification system. this combined respiratory gas will then be warmed and humidified and delivered to the patient via a nasal cannula. The total respiratory gas flow rate will be between 20-25 l/min, depending on participant´s preference. Then the oxygen fraction is adjusted until the subjects target oxygen saturation levels are achieved.
  Interventions: Device: Airvo humidifier
- Standard oxygen therapy (No Intervention): The control group will continue receiving the standard oxygen therapy prescribed by the department

INTERVENTIONS:
Device: Airvo humidifier — The Airvo humidifier has adjustable flow settings for delivery of fully saturated breathing gases at 37 °C, 100% humidity.
  Flow rates are adjustable between 15 and 45 l/min. Ambient air is drawn in by a low-capacity motor. When coupled to a medical oxygen supply, the regulation of delivered oxygen concentration is ensured.
  Arms: High Flow humidification system

SUMMARY:
The purpose of our study is to establish whether domiciliary use of the Airvo warm passover humidifier can reduce the number of exacerbations in patients with respiratory insufficiency. Participants must have a diagnosis of chronic obstructive pulmonary disease (COPD) and be in long term oxygen therapy (LTOT). The following questions will be investigated:

Do outpatients receiving long term oxygen therapy benefit if this is delivered through an Airvo humidification system. The proposed benefits under investigation are:

1. a reduction in the number of exacerbations and thus hospital admissions?
2. an increase in quality of life (QOL)?
3. an improved lung function and thus increased physical activity?

DETAILED DESCRIPTION:
Experience at Aalborg University Hospital's Department of Pulmonary Medicine (Lungemedicinsk Afdeling) in Denmark gives rise to a renewed interest in the investigation of the properties and effects of humidification in COPD patients in LTOT. For the last 5 years, the department has discharged fibrosis patients with oxygen flow > 6 l/min with a warm mist humidifier. The initiative has given clear indication that infection ratios can be reduced and the QOL increased. Many COPD patients experience improved oxygen saturation when oxygen treatment for respiration insufficiency is given with warm humidification.

Previous studies have typically concerned other patient categories and involved the use of cold-water humidifiers. To increase air moistening, the temperature must be raised as moisture absorption capability increases with temperature. The 2009 study of Rea et al. (9) examined the effect of warm humidification on COPD and bronchiectasis patients, who used a warm humidifier (MR 880) on average for two hours per day. LTOT was not an inclusion criterion in the study, and the severity of COPD varied. Despite the relatively short time of use the study demonstrated the beneficial effect of humidification on exacerbation frequency.

Our study therefore aims to examine the effect of using warm humidification as a minimum during the night - preferably for 8 hours.

In addition to their usual oxygen apparatuses, the treatment group will have an Airvo warm humidifier installed in the home. Their respiratory gas flow setting will be increased to 20-25 l/min based on patient preference; then the peripheral saturation readings will form the basis for adjusting the oxygen flow rate.

The control group will continue receiving the standard oxygen therapy prescribed by the department.

For the study to achieve the desired power, 190-200 patients across the two groups are required Appendix 3). Patients must have been diagnosed with severe/very severe COPD and be receiving long-term domiciliary oxygen treatment (LTOT)

For all participants, the following procedure will be adhered to:

1. Metrics at inclusion:

   * Demographic data
   * Pulmonary function measurement using spirometry
   * Exacerbations (by number of)

     * hospitalisation days in past year (data extracted from AS400)
     * antibiotics courses and prednisolone courses in past year (from prescription database)
     * exacerbations/self-treatment plans launched
   * 6-minute walk test
   * QOL measurement (St George's Respiratory Questionnaire)
   * Artery puncture (Airvo group only)
2. Metrics in project period at 1, 3, 6 and 9 months:

   Patients will be contacted by telephone on a date agreed in advance.
   * QOL measurement (St George's Respiratory Questionnaire). Form completed only after 6 months; sent to patient in advance.
   * Number of exacerbations/self-treatment plans launched
3. Metrics at project period completion (at 12 months):

Patients will be called in for an outpatient visit to the department

* Pulmonary function measurement (spirometry)
* St George's Respiratory Questionnaire (sent to patient prior to interview)
* 6-minute walk test
* Exacerbations in project period (by number of)

  * hospitalisation days in past year (data extracted from AS400)
  * antibiotics courses and prednisolone courses in past year (from prescription database)
  * exacerbations/self-treatment plans launched

Analysis and statistical processing of project data will be performed by statistician Hans Hockey of Biometricmatters Ltd, Hamilton, New Zealand. Power calculations based on anonymised data extracts from AS400 have already been performed.

Consultation with Mr Hockey has clarified that "events" and "visits" are synonymous terms. In the appendix the term "events" will be used, to indicate the number of contacts with the hospital.

According to Mr Hockey, risk time will be calculated as "the period of time for which a patient is at risk of the event being considered". Risk time thus corresponds to the time that the patient participates in the trial. The trial period is 12 months, but drop-out due to death or withdrawal for any other reasons is to be expected. All data will be included in the study, including data on dropouts.

This project protocol has been approved by the North Denmark Region scientific ethical committee (N-20110057).

ELIGIBILITY:
Inclusion Criteria:

* have severe/very severe COPD diagnosis
* have had chronic respiratory insufficiency for at least 3 months and be in steady oxygen therapy (LTOT) with a minimal supplement of 1 litre of oxygen per minute for at least 16 hours per day
* understand and accept oral and written information in Danish
* be capable of handling the Airvo warm humidifier after instruction.

Exclusion Criteria:

* Comorbidity (known malignant disease, terminal illness, dementia, uncontrolled mental illness)
* Bronchiectasis without simultaneous COPD diagnosis
* Treatment with BiPAP in the home
* Affected level of consciousness
* Smoking status change during project period.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-01; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Reduction in the number of exacerbations and thus hospital admissions, based on data on hospital admissions. | one year
  Outcomes relating to exacerbations will be recorded according to GOLD COPD guidelines:
  An exacerbation of COPD is defined as an event in the natural course of the disease characterized by a change in the patient's baseline dyspnea, cough and/or sputum that is beyond normal day-to-day variations, is acute in onset, and may warrant a change in regular medication in a patient with underlying COPD (3).
  At inclusion of the patient, the number of exacerbations (deterioration) in the last year, based on data on the need for antibiotics and/or prednisolone (corticosteroid), and hospital admissions will be registered. Data will be recorded via extracts from AS400 and the prescription database. To ensure data validity concerning redeemed prescriptions, patients will be asked about the number of self-treatment plans.
  At project completion, the same metrics are recorded for the entire period.

SECONDARY OUTCOMES:
increase in quality of life, measured by St George's Respiratory Questionnaire (SGRQ), | six month and one year
  All patients will be required to complete a health-related QOL questionnaire, the validated Danish version of the St George's Respiratory Questionnaire (SGRQ), see Appendix 1. Permission for use has been obtained from Professor Paul Jones, St George's University, London (Appendix 1).
  The questionnaire will be completed at inclusion, 6 months and 12 months.
improved lung function, using Spida 5 equipment. | one year
  The test will be performed by the project responsible nurse, or her deputy, using Spida 5 equipment. FEV1 and FEV1/FVC are recorded for both study groups. To ensure uniform measurement methods, the department's instructions on spirometry measurements will be followed
Improved physical ability, based on six-minute walk test. | one year
  The six-minute walk test, in which the patient walks as far as possible, will be used as a measure of functional work capacity. Patients will be encouraged to exert themselves. Any pauses will be included in the six minutes.
  To ensure uniform measurement methods, the department's instructions on spirometry measurements will be followed

CONTACTS AND LOCATIONS:
Overall Officials: Ulla M Weinreich, MD, Study Chair — Department for Pulmonary Medicine, Aalborg University Hospital, Denmark
Locations (1):
- Aalborg University Hospital, Aalborg, Nothern Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dansk Selskab for Almen Medicin. Klinisk vejledning: KOL i almen praksis - diagnostik, behandling, opfølgning, rehabilitering. 2008. Sundhedsstyrelsen: KOL - kronisk obstruktiv lungesygdom. Anbefalinger for tidlig opsporing, opfølgning, behandling og rehabilitering. 2007. Ringbæk, T, Taudorf, E, Overgaard, A, Sorknæs, A og Fabricius, P. Protokol for Iltbehandling i hjemmet. Dansk Lungemedicinsk Selskabs rekommandationer. 2006. Kampelmacher, MJ, Van Kesteren, RG, Alsbach, GPJ et al. Characteristics and complaints of patients prescribed long-term oxygen therapy in The Netherlands. Respiratory Medicine, 92, 70-75, 1998 Medicinsk Kompendium. Kap. 37 Lungesygdomme Cambell, EJ, Baker, MD, Crites-Silver, P. Subjective effects of humidification of oxygen for delivery by nasal cannula. A prospective study. Chest, 93, 289-293, 1988. Gorecka, D, Gorzelak, K, Sliwinski, P, Tobiasz, M, Zielinski, J. Effect of long term oxygen therapy on survival in patients with chronic obstructive pulmonary disease with moderate hypoxaemia. Thorax, 52, 674-679, 1997. Rea, H, McAuley, S, Jayaram, L, Garrett, J, Hockey, H et al. The clinical utility of long-term humidification therapy in chronic airway disease. Respiratory Medicine, 104, 525-533, 2010. Fisher & Paykel Healthcare. Airvo. Hospital Use Operating Manual. Siggaard-Andersen, O, Gøthgen, IH, Wimberley, PD, Fogh-Andersen, N. The oxygen status of the arterial blood revised: relevant oxygen parameters for monitoring the arterial oxygen availability. Scand J Clinical Lab Invest, 50, suppl. 203, 17-28, 1990.